CLINICAL TRIAL: NCT02225899
Title: Integration of Nutritional Metabolomics With Bioenergetics in Cystic Fibrosis
Brief Title: BioEnergetics and Metabolomics in Cystic Fibrosis
Acronym: BEAM-CF
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Alvarez, Assistant Professor, Emory University
Other Study IDs: IRB00073559; K01DK102851 (NIH)
Record Dates: First submitted 2014-08-21; First posted 2014-08-26 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect sputum, urine, and blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with Cystic Fibrosis: Cross-sectional, observational study
- healthy volunteers: Cross-sectional, observational study
- Subjects with CF in a vitamin D study: This is a longitudinal observational study in subjects enrolled in a high-dose vitamin D study. The investigator (Jessica Alvarez) does not assign the intervention to the subjects of the study.

SUMMARY:
With better medical care, patients with cystic fibrosis (CF), a life-threatening disease, are enjoying longer lives. As the CF life expectancy increases, conditions such as CF-related diabetes (CFRD) become more prevalent. Nutrition plays a major role in maintaining optimal health in cystic fibrosis (CF). This project is designed to investigate nutrition-related factors, such as diet and body composition, on outcomes in patients with CF. The data generated from this study will be used to inform future nutrition intervention studies in adults with CF and CFRD.

DETAILED DESCRIPTION:
Research methods include blood draws for plasma markers of oxidative stress and metabolomics (the measurement of thousands of small chemicals in the blood), magnetic resonance imaging (MRI, to assess energy capacity and thigh fat), dual energy X-ray absorptiometry (DEXA, to assess total and regional body fat and muscle), and indirect calorimetry (to assess resting energy expenditure and whole body fat oxidation). Clinically-relevant data, such as lung function, CF genotype, and diabetes status will be obtained from the electronic medical record and the CF Registry.

ELIGIBILITY:
Cystic Fibrosis

Inclusion Criteria:

* have confirmed CF diagnosis with at least one Class I to III CFTR mutations
* age ≥ 18 yrs
* on a clinically-stable medical regimen for 3 wks
* no intravenous or oral antibiotics for at least 3 wks prior to study visit

Exclusion Criteria:

* current pregnancy
* unwilling or unable to discontinue enteral tube feeds for one night before the study visit, if applicable
* most recent FEV1% <40%
* drug (recreational or prescription) or alcohol abuse
* pacemaker or any electronic implantable device
* unable to give informed consent

Healthy volunteers

Inclusion criteria:

* 18-50 yrs of age
* ambulatory status
* absence of hospitalization in the previous year except for accidents

Exclusion criteria:

* current pregnancy
* current active malignant neoplasm or history of malignancy (other than localized basal cell cancer of the skin) during the previous 5 years
* current respiratory disease including asthma, chronic obstructive pulmonary disorder, or emphysema
* current chronic autoimmune or pro-inflammatory disease
* history of tuberculosis, HIV, or other chronic infection
* previous diagnosis of type 1 or type 2 diabetes with active treatment with insulin or other glucose lowering medication
* advanced (≥ stage 3) renal disease
* body mass index (BMI) ≥ 30 kg/m2
* acute illness (such as a viral infection) within the past 2 weeks
* current use of any prescription medications that would indicate presence of an acute or chronic medical condition that may influence study results
* drug (recreational or prescription) or alcohol abuse
* weight instability (± 10% body weight within the last 6 months) or current participation in weight loss or weight gain program
* inability to provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with cystic fibrosis and healthy volunteers from the Atlanta community
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Acylcarnitine analysis by high-resolution liquid chromatography mass spectrometry | Baseline for cross-sectional study and 1 year for longitudinal study
  This will pe performed using targeted metabolomics methods

SECONDARY OUTCOMES:
quantitative plasma levels of specific plasma acylcarnitines | Baseline for cross-sectional study and 1 year for longitudinal study
  This will be measured in fasted blood

OTHER OUTCOMES:
whole-body fasting fat oxidation | Baseline for cross-sectional study and 1 year for longitudinal study
  This will be assessed using indirect calorimetry
31P-magnetic resonance spectroscopy (MRS)-derived measures of resting thigh skeletal muscle bioenergetic metabolism | Baseline for cross-sectional study
  This will be assessed using MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Alvarez, PhD, RD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States